CLINICAL TRIAL: NCT02856100
Title: Comparison of PSMA-based 18F-DCFPyL PET/CT to Conventional Imaging in the Evaluation of Patients With Castration-Resistant Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: J15232; IRB00082289 (Other: JHMIRB)
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with CRPC, evidence of metastases, planned treatment
  Interventions: Drug: 18F DCFPyL- Radiopharmaceutical

INTERVENTIONS:
Drug: 18F DCFPyL- Radiopharmaceutical

SUMMARY:
We intend to validate 18F-DCFPyL for imaging patients with metastatic, castrate-resistant PCa (CRPC), so that it may be used to full advantage in supporting existing and emerging therapies for a spectrum of patients suffering from PCa. In this study we will image patients with CRPC undergoing second-line anti-androgen therapy (enzalutamide or abiraterone) using 18F-DCFPyL-PET/CT for detection of metastases and therapeutic monitoring, with correlation to standard-of-care conventional imaging modalities (CIM) (CT, bone scan) and clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years and male
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Patients starting abiraterone (but naïve to enzalutamide) or starting enzalutamide (but naïve to abiraterone)
* Prior docetaxel-based chemotherapy is permitted but not required
* Documented metastatic prostate cancer progression as assessed by the treating oncologist with either one or both of the following:

  * Rising PSA over a minimum 1-week interval
  * Radiographic progression in soft tissue and/or bone
* Ongoing androgen deprivation with serum testosterone < 50 ng/dL (< 1.7 nM)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Hemoglobin ≥ 90 g/L independent of transfusion
* Platelet count ≥ 100,000/μL
* Serum albumin ≥ 30 g/L
* Serum creatinine < 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min
* Serum potassium ≥ 3.5 mmol/L

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Abnormal liver functions consisting of any of the following:

  * Serum bilirubin ≥ 1.5 x ULN (except for patients with documented Gilbert's disease)
  * AST or ALT ≥ 2.5 x ULN, (for patients with known liver metastasis, AST or ALT ≤ 5 x ULN is allowed)
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg)
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 12 months
* Known brain metastasis
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of orally administered hormonal agents.
* Acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a NCI CTCAE (version 4.0) grade of ≤ 1; chemotherapy-induced alopecia and grade 2 peripheral neuropathy are allowed
* Current enrollment in an investigational drug or device study, or participation in such a study within 30 days of first administration of the hormonal agent.
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study
* Not willing to comply with the procedural requirements of this protocol
* Patients who have partners of childbearing potential who are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRPC and planned treatment with evidence of metastases on conventional imaging modality (CIM) (CT and/or bone scan)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in number of metastatic lesions detected on 18F-DCFPyL PET/CT | up to 2 years
  Change in number of metastatic lesions detected from baseline standard of care conventional imaging (CT and Bone Scan) to 18F-DCFPyL PET/CT at 8-12 weeks post- anti-androgen therapy (standard of care)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States